CLINICAL TRIAL: NCT03463356
Title: The Development and Evaluation of a Brief Shame Intervention Module: Proof of Concept in Social Anxiety Disorder
Brief Title: Brief Shame Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Miami University (Other)
Responsible Party: Principal Investigator, Elise Clerkin, Associate Professor, Miami University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01474r
Record Dates: First submitted 2018-03-01; First posted 2018-03-13 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Shame; Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Intervention Model Description: non-concurrent multiple baseline design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Shame Intervention (Experimental): Participants will complete a two shame intervention sessions approximately one week apart.
  Interventions: Behavioral: Shame Intervention

INTERVENTIONS:
Behavioral: Shame Intervention — In the Shame Intervention, participants will meet with a therapist and learn to: 1) Recognize the experience of shame, 2) Understand the connection between shame and social anxiety, 3) Identify shame triggers and vulnerabilities, 4) Identify the thoughts and behaviors that keep participants stuck in shame, and 5) Learn how to use new, healthier thoughts and behaviors that will help participants move through and decrease shame.

SUMMARY:
The current project will develop and test a brief 2-session shame intervention in individuals diagnosed with social anxiety disorder (SAD). Using a non-concurrent multiple baseline design, the investigators will determine whether the brief shame intervention leads to reductions in trait self-reported shame and state shame in response to an in vivo stressor task. The investigators will also evaluate the effect of changes in shame on trait SAD symptoms.

ELIGIBILITY:
Inclusion Criteria:

-≥ 18 years old

* fluent in English, in terms of verbal and written competence
* meet diagnostic criteria for social anxiety disorder (as assessed by the Diagnostic Interview for Anxiety, Mood, and OCD and Related Neuropsychiatric Disorders; Tolin et al., 2016)
* have elevated levels of shame (i.e., score 1 SD above the Test of Self-Conscious Affect-3 [TOSCA-3] means reported by an unselected undergraduate sample [M = 33.62, SD = 8.64])
* endorse a desire to decrease their levels of shame and/or social anxiety.

Exclusion Criteria:

* currently receiving cognitive-behavioral therapy specifically for social anxiety or shame
* have begun taking or had a change in dosage of psychotropic medication in the past six weeks
* do not achieve baseline stability

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Test of Self-Conscious Affect-3-Short Form | Participants indicate likelihood of responses to scenarios. Administered at B1-B5 and T1-T5. B1-B5 occur ~1 week apart. T1 occurs ~1 week after the final baseline. T1-T4 each occur within ~2 weeks of each other. T5 occuring ~1 month after T4.
  Self-report of how likely an individual is to react to 11 scenarios with shame responses

SECONDARY OUTCOMES:
Change in Liebowitz Social Anxiety-Self-Report | Participants report on symptoms during the past week. Administered at T1-T5. T1-T4 each occur within ~2 weeks of each other. T5 occurs ~1 month after T4.
  Self-report of social anxiety symptoms
Change in Brief State Anxiety Measure | Participants report on symptoms experienced during the speech task. Administered at T1 and T4. T4 occurs within ~6 weeks after T1.
  Self-report of levels of anxiety experienced during the speech task
Change in Shame Inventory | Participants report on typical experience of symptoms. Administered at T1, T4, and T5. T4 occurs within ~6 weeks after T1. T5 occurs ~1 month after T4.
  Self-report of shame symptoms
Change in State Shame and Guilt Measure | Participants report on symptoms experienced during the speech task. Administered at T1 and T4. T4 occurs within ~6 weeks after T1.
  Self-report of levels of shame experienced during the speech task

OTHER OUTCOMES:
Change in Center for Epidemiologic Studies Depression Measure | Participants report on symptoms experienced during the past week. Administered at T1, T4, and T5. T4 occurs within ~6 weeks after T1. T5 occurs ~1 month after T4.
  Self-report measure of depressive symptoms
Change in Clinical Perfectionism Measure | Participants report on symptoms experienced during the past month. Administered at T1, T4, and T5. T4 occurs within ~6 weeks after T1. T5 occurs ~1 month after T4.
  Self-report measure of perfectionism
Change in Eating Disorder Inventory - 3rd Version | Participants report on typical experience of symptoms. Administered at T1, T4, and T5. T4 occurs within ~6 weeks after T1. T5 occurs ~1 month after T4.
  Self-report measure of eating disorder symptoms
Change in Brief Fear of Negative Evaluation Measure-II | Participants report on typical experience of symptoms. Administered at T1, T4, and T5. T4 occurs within ~6 weeks after T1. T5 occurs ~1 month after T4.
  Self-report measure of fear of negative evaluation
Change in Self Beliefs about Social Anxiety | Participants report on typical experience of symptoms. Administered at T1, T4, and T5. T4 occurs within ~6 weeks after T1. T5 occurs ~1 month after T4.
  Self-report measure of social anxiety disorder relevant maladaptive beliefs

CONTACTS AND LOCATIONS:
Overall Officials: Marie Parsons, M.A., Principal Investigator — Miami University
Locations (1):
- Anxiety Cognition and Emotion Laboratory, Oxford, Ohio, United States

IPD SHARING:
Plan to Share IPD: No